CLINICAL TRIAL: NCT04944056
Title: Effect of Compression Mobilization (Kaltenborn Technique) in Knee Osteoarthritis Patients
Brief Title: Effects of Compression Mobilization in OA Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mir Arif Hussain (Industry)
Responsible Party: Sponsor-Investigator, Mir Arif Hussain, Research Head, Aqua Medical Services (Pvt) Ltd
Organization: Aqua Medical Services (Pvt) Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shakeeba Shahzadi 00189
Record Dates: First submitted 2021-06-22; First posted 2021-06-29 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Osteo Arthritis Knee
Keywords: NPRS, mBBS, MMT, O.A

STUDY DESIGN:
Intervention Model Description: The experimental Group received compression mobilization with Conventional Physiotherapy and the control group received Conventional Physiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): It includes ultrasound therapy, glides, exercises and home plan.
  Interventions: Other: conventional physiotherapy
- Experimental Group (Experimental): It includes ultrasound therapy, glides, exercises, compression mobilization and home plan.
  Interventions: Other: compression mobilization

INTERVENTIONS:
Other: conventional physiotherapy — * Ultrasound therapy 3-4 minutes.
  * Tibiofemoral AP and PA glides 1 set x10reps x 3 sets.
  * Patellar glides 1 set x 5 reps x 3 sets.
  * Quads isometrics 1 set x 10 reps.
  * Hams self stretching 1 sets x 10 reps.
  Home plan:
  * Quads isometrics 1 set x 10 reps.
  * Hams self stretching 1 sets x 10 reps.
  * Active range of motion.
  Arms: Control Group
Other: compression mobilization — * Ultrasound therapy 3-4 minutes.
  * Tibiofemoral AP and PA glides 1 set x10reps x 3 sets.
  * Patellar glides 1 set x 5 reps x 3 sets.
  * Quads isometrics 1 set x 10 reps.
  * Hams self stretching 1 sets x 10 reps.
  * Compression mobilization 1 set x 10 reps x 3sets.
  Home plan:
  * Quads isometrics 1 set x 10 reps.
  * Hams self stretching 1 sets x 10 reps.
  * Active range of motion.
  Arms: Experimental Group

SUMMARY:
The study Design was randomized control trial in which data was collected From Riphah Rehabilitation And Research Center and Pakistan Railway Hospital-IIMCT. Convenient sampling technique was used for data collection. 39 patients having knee osteoarthritis were recruited in this study. After taking consent from patients, patients were divided randomly into two groups through lottery method. The Experimental Group received compression mobilization with Conventional Physiotherapy (n = 19) and the Control group received Conventional Physiotherapy (n = 20). Research data was collected through structural questionnaire. the main variables were ROM, MMT, Muscle length and mBBS.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a disease which since long times is considered to be a "wear and tear" malfunctioning disease leading to a loss of cartilage. Osteoarthritis is considered as a "degenerative joint disease Osteoarthritis is a term used for disease in which destruction of cartilage is involved (articular), with a bone thickening (subchondral) and formation of new bone. . Joint swelling is also considered as one significant clinical feature of osteoarthritis attributes to inflammation. Osteoarthritis is one of the most common type in arthritis as well as the major cause of chronic musculoskeletal pain. In addition it is attributed to mobility disability in the elder or high aged population all over the world. If we have a glimpse of Asia, prevalence rate of knee osteoarthritis is believed to be higher in the elder population most probably in women. Susan et all conducted a mega level study related to symptomatic OA, where it has been observed that there is an increasing shift in the incidental rates of OA with the age. So, it was concluded that incidence related to knee OA in women limiting the age between 70-89, approached per year is 1% in women and they had the higher rates as compared to males, especially once they are over 50 years of age. Levelling-off or declining shift tends to occur for both groups approximately at the age of 80. Research says that in China, this prevailing rate of mentioned osteoarthritis disease is 7.50%, with a ratio of 10.9 & 13.6% in males and females respectively. Bangladesh and India reports 5.80 & 10.20% respectively. Now considering mainland of Pakistan, 28% urban whereas 25% rural population suffer this particular disease.

Women are likely to suffer more with the OA as compared to men and they also tend to undergo the disease of OA with more severity. The marked increase of OA in females at menopause stages has directed towards investigational hypothesis that hormonal imbalance factor may perform a significant role for the developing of OA. However, results appearing on estrogen effects, either it's endogenous or exogenous, on OA as revealed from various observational researches have been contradictory. In a randomize clinical trials(the Heart and Estrogen/Progestin Replacement Study) considering the group of elder postmenopausal females suffering from heart disease, none significant variation was observed in persistence of knee pain or any associated disability while comparing those undergoing estrogen plus progestin therapy or those taking placebo.

The prevalence of OA disease and joints patterns that are effected by OA possibly vary amongst the ethnic and racial groups. The frequency of Hand and Hip OA was found remarkably less in Chinese, concluded in the Beijing Osteoarthritis Study, in resemblance to whites researched under Framingham Study. it's important to mention that Chinese females observed under the Beijing Osteoarthritis Study had considerably high prevalence of both symptomatic knee OA and radiographic knee OA as compared to white females at Framingham Study. Results while having consideration of Johnston County Osteoarthritis Project have showed the prevalence of hip OA in African American females(23%) was similar to that in white ladies (22%), with a conclusion that prevalence was a bit higher in African American men (21%) than that in white.

Result of various studies showed that dietary factor is a subject of considerable interest related to OA affected individuals. Vitamin D is considered as most advantageous nutritional factor for OA patients. Insufficiency of this specified vitamin will lead to bones thinness, brittleness or any mishaps.

Corpulence (Obesity leading to overweight) have since long been predicted as the most potent risk factor to OA, especially knee OA. A more consistence and reliable evidence found is that the alarming effects occurs due to obesity are the risks of bi-lateral radiography and symptomatic hip OA. So, it is considered that application of increased loads on joints is probably a major cause, but not necessarily, a mechanism by which the obesity results into hip or knee OA. Whereas, an application of overloading the knee and hip joints could possibly directed towards synovial joint breakdown and failure of ligamentous as well as other structural support.

A lot many studies provides evidence that knee injury is surely one of the strongest factor for risking OA. Severe conditions of injury to joints structures, particularly mentioning the meniscal tear that requiring meniscectomy, or trans-articular fracture or anterior cruciate ligament injury; may these all results into increased risk involvement of OA development and also musculoskeletal symptomatology.

Repeated use of particular joints for work is marked with the increasing risk of OA. The risk factor involved in the development of knee OA was at least two times more for men whose consistency in jobs require both kneeling and carrying or squatness in a mid-life would definitely have more risk of developing OA by the nature of their commitments as compared to women whose job commitments do not offer these physical activities in common. Therefore, its a must mention that knee OA risks which are associated with squatness or kneeling are much higher amongst those who are overweighed or who are indulgent in lifting.

ELIGIBILITY:
Inclusion Criteria:

* Age Limit 30 to 60
* Unilateral OA Knee
* Moderate OA

Exclusion Criteria:

* No Associated Bone Disease
* Lumber Radiculopathy
* Osteoporosis
* Any MSK Deformity

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-07-11 (Actual); Study Completion 2021-07-11 (Actual)

PRIMARY OUTCOMES:
Vernier Calliper For Joint Gap Measurement. | 2 weeks
  Vernier caliper, instrument for making very accurate linear measurements introduced in 1631 by Pierre Vernier of France. It can be used for joint space via x-ray radiograph of a joint.
Numeric Pain Rating Scale | 2 weeks
  Numeric pain rating scale is a scale used to quantify pain intensity. It is divided into eleven equal parts; for example 0 - 10. O means that there is no pain at all, 1 - 3 divisional range falls in the mild category pain , 4 - 6 indicates the symptoms of moderate pain while 7 - 10 reading symptoms the severity of pain.
Goniometry for knee ROM | 2 weeks
  The Range of motion was assessed by Goniometer. The placement of goniometer for flexion as follows the Axis of goniometer was placed at lateral epicondyle of femur laterally , stationary arm was along femur and the moving arm was along the fibula and the patient position was supine then ask the patient to flex knee until hip flexion came up to 90 degrees while monitors the measurements through goniometer .
Modified Berg Balance tool | 2 weeks
  The Berg Balance Scale (BBS) is based on 14 items common to daily life activities used to evaluate functional balance .here berg balance scale is used to assess patients proprioception through different tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Shakeeba Shahzadi, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation And Research Center and Pakistan Railway Hospital-IIMCT, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berenbaum F. Osteoarthritis as an inflammatory disease (osteoarthritis is not osteoarthrosis!). Osteoarthritis Cartilage. 2013 Jan;21(1):16-21. doi: 10.1016/j.joca.2012.11.012. Epub 2012 Nov 27. PMID 23194896
- [Background] Blagojevic M, Jinks C, Jeffery A, Jordan KP. Risk factors for onset of osteoarthritis of the knee in older adults: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2010 Jan;18(1):24-33. doi: 10.1016/j.joca.2009.08.010. Epub 2009 Sep 2. PMID 19751691
- [Background] Brandt KD, Fife RS, Braunstein EM, Katz B. Radiographic grading of the severity of knee osteoarthritis: relation of the Kellgren and Lawrence grade to a grade based on joint space narrowing, and correlation with arthroscopic evidence of articular cartilage degeneration. Arthritis Rheum. 1991 Nov;34(11):1381-6. doi: 10.1002/art.1780341106. PMID 1953815
- [Background] van Saase JL, van Romunde LK, Cats A, Vandenbroucke JP, Valkenburg HA. Epidemiology of osteoarthritis: Zoetermeer survey. Comparison of radiological osteoarthritis in a Dutch population with that in 10 other populations. Ann Rheum Dis. 1989 Apr;48(4):271-80. doi: 10.1136/ard.48.4.271. PMID 2712610
- [Background] Rhon D. Re: Zhang W, Moskowitz RW, Nuki G, et al. OARSI recommendations for the management of hip and knee osteoarthritis, Part II: OARSI evidence-based, expert consensus guidelines. Osteoarthritis Cartilage 2008;16:137-62. Osteoarthritis Cartilage. 2008 Dec;16(12):1585; author reply 1589. doi: 10.1016/j.joca.2008.04.019. Epub 2008 Jun 2. No abstract available. PMID 18515155
- [Background] Heidari B. Knee osteoarthritis prevalence, risk factors, pathogenesis and features: Part I. Caspian J Intern Med. 2011 Spring;2(2):205-12. PMID 24024017
- [Background] Fransen M, Bridgett L, March L, Hoy D, Penserga E, Brooks P. The epidemiology of osteoarthritis in Asia. Int J Rheum Dis. 2011 May;14(2):113-21. doi: 10.1111/j.1756-185X.2011.01608.x. PMID 21518309
- [Background] Zhang Y, Niu J, Kelly-Hayes M, Chaisson CE, Aliabadi P, Felson DT. Prevalence of symptomatic hand osteoarthritis and its impact on functional status among the elderly: The Framingham Study. Am J Epidemiol. 2002 Dec 1;156(11):1021-7. doi: 10.1093/aje/kwf141. PMID 12446258
- [Background] Haq SA, Darmawan J, Islam MN, Uddin MZ, Das BB, Rahman F, Chowdhury MA, Alam MN, Mahmud TA, Chowdhury MR, Tahir M. Prevalence of rheumatic diseases and associated outcomes in rural and urban communities in Bangladesh: a COPCORD study. J Rheumatol. 2005 Feb;32(2):348-53. PMID 15693098
- [Background] Nelson AE, Braga L, Renner JB, Atashili J, Woodard J, Hochberg MC, Helmick CG, Jordan JM. Characterization of individual radiographic features of hip osteoarthritis in African American and White women and men: the Johnston County Osteoarthritis Project. Arthritis Care Res (Hoboken). 2010 Feb;62(2):190-7. doi: 10.1002/acr.20067. PMID 20191517
- [Background] Kon E, Mandelbaum B, Buda R, Filardo G, Delcogliano M, Timoncini A, Fornasari PM, Giannini S, Marcacci M. Platelet-rich plasma intra-articular injection versus hyaluronic acid viscosupplementation as treatments for cartilage pathology: from early degeneration to osteoarthritis. Arthroscopy. 2011 Nov;27(11):1490-501. doi: 10.1016/j.arthro.2011.05.011. Epub 2011 Aug 10. PMID 21831567
- [Background] Takasaki H, Hall T, Jull G. Immediate and short-term effects of Mulligan's mobilization with movement on knee pain and disability associated with knee osteoarthritis--a prospective case series. Physiother Theory Pract. 2013 Feb;29(2):87-95. doi: 10.3109/09593985.2012.702854. Epub 2012 Jul 30. PMID 22844980